CLINICAL TRIAL: NCT03332121
Title: Phase Ia Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of Recombinant Humanized Anti-CD20 Monoclonal Antibody for Injection(B001)
Brief Title: B001 in Patients With CD20 Positive B-cell Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B001-101
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: CD20 Positive B Cell Non-Hodgkin's Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B001,B001 dose escalation (Experimental): 5 groups with different dose: 350mg/700mg/1000mg/1500mg/2000mg
  Interventions: Biological: B001

INTERVENTIONS:
Biological: B001 — 4 times intravenous injection totally,dosing at Day1,Day35,Day56,Day77

SUMMARY:
It's the first-in-human study of Recombinant Humanized Anti-CD20 Monoclonal Antibody for Injection (B001). The main purpose of this study is to explore the safety and tolerance of B001 for patients with CD20 positive B-cell non Hodgkin's lymphoma. It will also explore the PK/PD manner and ORR in this study.

DETAILED DESCRIPTION:
Phase I dose escalation study

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75, male or female.
2. Patients with the following histologically-documented hematologic malignancy: CD20 positive B-cell non Hodgkin's lymphoma (NHL) or chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), according to 2016 WHO Classification of Lymphoma.
3. Patients with relapsed/refractory CD20 positive B cell NHL (including CLL/SLL )
4. Life expectancy of at least 6 months.
5. ECOG-PS score of 0-1.
6. For patients of reproductive potential, pregnancy test should be negative 7 days before treatment , and use of a reliable means of contraception during the study and 12months after discontinuing treatment. Males should be willing to use barrier contraception during the study and 12months after discontinuing treatment.
7. Provision of signed and dated ,written informed consent prior to any study specific procedures, sampling and analyses.

Exclusion Criteria:

1. Serious blood, renal or hepatic function impairment:

   * Absolute neutrophil count(ANC)<1.0*10^9/L（Except for those with bone marrow invasion）
   * Lymphocyte Count(LYM)>50*10^9/L
   * Haemoglobin(Hb)<70g/L（Except for those with bone marrow invasion）
   * Platelet count(PLT)<50*10^9/L（Except for those with bone marrow invasion）
   * Creatinine (Cr)>1.5xULN
   * Alanine transaminase (ALT)or Aspartate aminotransferase(AST)>2.5xULN
   * Total bilirubin (TBIL)>2xULN
2. Patients with any anti-tumor treatment (including steroid treatment) within 4 weeks or with any chronic unresolved toxicities from prior therapy greater than Grade 2 according to NCI-CTCAE 4.03.
3. Rituximab or any other anti-CD20 monoclonal antibody treatment within 3 weeks.
4. received blood transfusion and hemopoietic stimulating factor,eg. colony-stimulating factor (CSF)、Erythropoietin(EPO) within 2 weeks.
5. Radiotherapy within 3 months.
6. Major surgery within 28 days
7. History of tumor vaccine treatment.
8. Live-virus (live attenuated) vaccine treatment within 28 days
9. High dose of steroid treatment (hydroprednisone >10mg/day or relevant dose of other drugs)
10. Patients with history of hematopoietic stem cell transplantation or planning to receive hematopoietic stem cell transplantation within 3 months.
11. Patients with history of Gastrointestinal perforation and/or fistula within 6 months.
12. Lymphoma in CNS, ADIS related lymphoma
13. Active infection by bacteria,virus,fungus which required hospitalization or severe infection required intravenous administration of antibiotics
14. Concomitant severe disease including but not limited to:

    * Known HIV or ADIS related disease
    * Asthma or interstitial lung disease or severe COPD
    * Myocardial infarction, unstable angina, Cardiovascular interventional surgery, Congestive heart failure(CHF; NYHA Grade II-IV), symptomatic or poorly controlled arrhythmia within 6 months before enrolling
    * The systolic pressure ≥140mmHg,or diastolic pressure≥90mmHg post treatment.
    * Acute or chronic hypotension(<90/60mmHg)
    * History of toxic epidermal necrolysis or Stevens-Johnson syndrome
    * Rheumatoid arthritis Granulomatous angiitis or microscopic polyangiitis
    * Ileus or history of following disease: inflammatory bowel disease or extensive intestinal resection(extensive bowel resection or hemicolectomy, combining chronic diarrhea), Crohn's disease, ulcerative colitis or chronic diarrhea.
    * Previous or concomitant malignant, except basal-cell carcinoma or squamous cell carcinoma and/or cervical carcinoma in situ or effectively treated hematological malignancy and solid tumor that has been remission for more than 3 years and is considered to be cured.
    * Any history may affect the study result: increasing dosing risk or affect lab values and Judgment by the investigator that the patient should not participate in the study,
15. HBsAg positive; HBcAb positive and HBV-DNA≥upper limit of detection, HCV positive; HIV positive
16. Allergy to humanized antibody or human-mouse chimeric antibody.
17. Woman who are breast feeding or pregnant
18. Judgment by the investigator that the patient should not participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Safety of B001 as assessed by adverse reactions and events | 42 days
  Incidence and intensity of adverse events according to NCI CTCAE 4.03 associated with increasing doses of B001

SECONDARY OUTCOMES:
Concentration-time curve of B001 | 112 days
  Measure the concentration of B001 in serum at different time point to get a concentration-time curve.
PD results of B001 | 112 days
  Measure the number of CD19 positive B cell in peripheral blood
Immunogenicity of B001 | 112 days
  Content analysis of anti-B001 antibody
ORR of B001 | 112 days
  Objective response rate according to Response Criteria for Lymphoma（not including PET）and CLL Response Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Doctor, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Junyuan Qi, Doctor, Principal Investigator — Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (2):
- China (2):
  - The second affiliated hospital of Guangzhou medical university, Guangzhou, Guangdong
  - Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality